CLINICAL TRIAL: NCT05305391
Title: Low-grade Inflammation and Gut Symptoms From A2 and Hydrolyses A1 Milk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Kaisa Linderborg, Principal Investigator, University of Turku
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: MILK3
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Milk Intolerance
MeSH Terms: conditions — Lactose Intolerance | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A2 milk + placebo (Experimental): A2 whole milk, 3.5% fat, heat-treated; placebo capsule without enzyme
  Interventions: Other: Dietary intervention
- A2 milk+ lactase enzyme (Experimental): A2 whole milk, 3.5% fat, heat-treated; lactase capsule
  Interventions: Other: Dietary intervention
- Protein-hydrolyzed A1 milk + placebo (Experimental): Protein-hydrolyzed lactose-free milk, 3% fat, heat-treated; placebo capsule without enzyme
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — The arising gastrointestinal symptoms and inflammation markers from consumption of milk + lactase capsule / placebo.

SUMMARY:
The aim of this study is to reveal how different forms of milk casein, lactose and moderate breakdown of proteins affect the symptoms that may arise from milk and markers of inflammation in volunteers receiving symptoms from milk. Research hypotheses are: 1) Protein hydrolyzed milk is as tolerated or better tolerated than A2 milk, and 2) Lactose is the main causative agent of stomach symptoms in milk-sensitive individuals.

ELIGIBILITY:
Inclusion Criteria:

* Perceive disturbing gut symptoms from regular milk
* Commits to the research diet for the whole research period
* Age: 18-65
* BMI: 18.5-30
* Healthy (normal kidney, liver and thyroid function and self-reported)

Exclusion Criteria:

* Milk allergy
* Regular medication (other than contraceptives) or medication affecting the gut
* Recent course of antibiotics (< 3 months prior the study)
* Pregnancy or lactation
* Diagnosed bowel disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal symptoms | day 0 - day 3
  Gastrointestinal symptoms (self-reported) as measured by a questionnaire. The questionnaire is divided into seven types of gastrointestinal discomfort, and also includes a possibility to describe a gastrointestinal discomfort outside these seven given alternatives. The severity of the symptoms is self-reported on a three-step scale.
Inflammation markers | day 4
  Differences in inflammation markers (from plasma) are measured as a baseline before the study and then after each study arm.
Calpro | day 4
  Faecal calprotectin (from faecal sample) is used to measure inflammation status of the gut.
Stool quality and defecation regularity | day 0 - day 3
  Stool quality and defecation regularity are self-reported with Bristol scale during the consumption of milks.

CONTACTS AND LOCATIONS:
Locations (1):
- Food Chemistry and Food Development, Department of Life Technologies, University of Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: No